CLINICAL TRIAL: NCT00357799
Title: VeinViewer for Peripheral IV Placement in Children With Difficult IV Access
Brief Title: VeinViewer for Peripheral IV Placement in Children With Difficult Intravenous (IV) Access
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital and Health System Foundation, Wisconsin (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, Kenneth Yen, Associate Professor of Pediatrics (Emergency Medicine) and Population Health (Epidemiology), Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHW 06/139, GC 185
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Catheterization, Peripheral; Phlebotomy
Keywords: Venipuncture; Randomized Controlled Trial; Intravenous Access; Children; Emergency Department Nursing; VeinViewer; Pediatrics; Emergency Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VeinViewer Arm (Active Comparator): Attempts at IV placement will be made with use of the VeinViewer Machine
  Interventions: Device: VeinViewer
- Conventional Method (No Intervention): IV attempted with conventional method

INTERVENTIONS:
Device: VeinViewer — Using the VeinViewer, IV attempts will be made
  Arms: VeinViewer Arm

SUMMARY:
Hypothesis: The first attempt success rate for peripheral IV insertion for children with difficult IV access (difficult IV access [DIVA] score ≥ 4) by nurses using the VeinViewer guided technique is better than conventional method of IV placement.

Specific Aims:

1. To investigate if use of the VeinViewer can improve the success of peripheral IV placement in children with difficult IV access
2. To validate the DIVA score

Design: Prospective randomized controlled trial/Convenience sample

Subjects: Children (0-18) presenting to the emergency department who require an IV as determined by examining physician and with a DIVA score ≥ 3 during times when VeinViewer machine is available and a VeinViewer trained participating nurse is on duty.

Variables:

Outcome Variables: First IV attempt success rate

Predictor Variables: IV technique used, other potential modifiers (age, weight, height, skin shade, indication for IV, history of prematurity and, vein visibility/palpability after tourniquet)

Methods: Subjects who meet inclusion criteria will be randomized to either conventional IV technique or VeinViewer guided technique. The nurse will attempt the IV depending on the randomization. Success or failure on first IV attempt will be recorded. If unsuccessful, other attempts will be tried until a successful IV is placed or the physician decides to give an alternative therapy that does not need IV access.

Statistics: A chi square test will be used to compare the proportion of subjects with successful first attempt IV placement using the VeinViewer technique to that using the conventional method with 95% confidence interval. We, the researchers, will look at the median number of attempts to place an IV in each of the groups. Logistic regression will be performed to test for independent associations. Information collected during the study will also be used for validation of the DIVA score.

Risks: No extra risks are expected above that of receiving a standard IV. The standard risk of bleeding, bruising, pain, and infection will be possible regardless of technique used. The VeinViewer does not expose the patient the ionizing radiation. The use of the VeinViewer technique may increase the time need to place an IV in.

Potential Benefits: With this study, we, the researchers, hope to improve the success rate of children with difficult IV placement in the Emergency Department.

DETAILED DESCRIPTION:
Introduction:

Attempting to get peripheral intravenous (IV) access can be one of the most frustrating and irksome tasks medical professionals encounter. Many medical therapies require the placement of an IV. In an emergency situation, it can be the lifeline that makes the difference between a good or bad outcome. Determinants of successful IV placement include the skill and expertise of the person who places the IV, the veins of the person who receives the IV, and luck.

These difficulties are often magnified in children. Children have smaller veins. Children come in different sizes and shapes. Children are often uncooperative. Not uncommonly, multiple attempts at IV placement are required before success. The more attempts that are needed to get an IV placed, the more pain and anxiety a child experiences. Getting an IV in a timely manner can alter parental perceptions of the quality of care and improve parental satisfaction. Developing methods to improve success rate of IV placement has obvious benefits.

During a previous study, we were able to demonstrate that in 25% of the patients in our pediatric emergency department who have an IV placement attempt will fail the first IV attempt. We were able to develop a scoring system (termed DIVA score) that we believe will aid in identifying those more likely to have a failed first IV attempt and so therefore may more likely benefit from our intervention (VeinViewer™). By attempting to demonstrate improved success on those with an increase likelihood of failure on first IV attempt, we believe that we will decrease the number of subjects needed to show an effect and to limit this potentially resource intensive technique to those most likely to benefit.

The VeinViewer™ is an infrared imaging system that utilizes near-infrared light and other technologies to project a real-time image of the location and orientation (up to 0.06mm) of veins onto the surface of patient's skin. The VeinViewer™ received FDA clearance in August 2004 as a class I device. The VeinViewer's Infrared Light is considered harmless. We believe a potential application for the VeinViewer™ is to improve the success rate of IV insertion in

Objectives:

1. To investigate if use of the VeinViewer™ can improve the success of peripheral IV placement in children with difficult IV access (DIVA score ≥ 3).
2. To validate the DIVA (difficult IV access) score

Hypothesis:

1. The first stick success rate for peripheral IV insertion for children with difficult IV access in a pediatric emergency department (DIVA score ≥ 3) by registered nurses using VeinViewer™ guided technique is better than conventional method of IV placement.
2. The DIVA score is a valid scoring system to identify those who are more likely to have failed first IV attempt.

Methods:

Study Design: Prospective randomized controlled trial.

Randomization: Subjects will be randomized to either get the VeinViewer™ technique or the conventional method. Serially number sealed opaque study packets with the blocked randomization will be created.

Subjects:

Inclusion criteria:

* Presentation to the ED at the CHW
* 0 to 19 years of age
* Requires a peripheral IV as determined by the examining physician
* DIVA score ≥ 3 (a clinical scoring system that identifying difficult IV access that gives 2 points for vein not visible after tourniquet, 2 for vein not palpable after tourniquet, 1 for age 1-2yo, 3 for age < 1 yo, 3 for history of prematurity)
* During times when VeinViewer™ machine and participating nurse is available

Exclusion criteria:

* Central line available
* Immunocompromised patient
* Requirement for immediate IV placement (Patient's condition would potentially be compromised if there is a time delay in IV placement.)

Patients who present to the emergency department and whom an IV is ordered will be screened for inclusion in the study by research assistants, nursing, or investigators. A DIVA score will be determined. Those with a score ≥ 3 will be approached to take part in the study. Informed parental consent will be obtained. Patient assent will be obtained for children 7 years of age and older).

Measurements:

Predictor Variables: VeinViewer™ or conventional methods

Main Outcome Variable: Success or failure of peripheral IV placement on first attempt

Secondary Outcome Variable: Number of attempts to successful IV placement

Data to be collected (potential modifiers for successful IV placement):

* Age (Date of Birth)
* Number of IV attempts until success or quitting
* Date of visit
* Location of IV attempts
* Weight
* Reason for IV (Fluid, medication, other)
* Height
* Dermablend skin color category
* History of prematurity
* Pre-attempt analgesia used
* Vein visibility after tourniquet
* Vein palpability after tourniquet
* Technique used (VeinViewer™/Conventional technique)

Conventional method:

A tourniquet is applied. The nurse identifies a target vein visually and tactilely in one of several areas of possible IV sites (dorsum of the hand, antecubital fossa, or forearm). The area is cleaned with an alcohol pad. The nurse then inserts an 18-24 gauge IV needle/catheter and looks for a flashback. The tourniquet is released. The IV is then flushed. If the IV flushes well, then the IV is secured in the usual manner. A secured flushed IV is the definition of a successful IV placement.

VeinViewer™ technique:

A tourniquet is applied. Using the VeinViewer™ the nurse identifies a vein for cannulation. A tourniquet is applied. The nurse then attempts to insert an 18-24 gauge IV needle/catheter and looks for a flashback. The tourniquet is released. The IV is then flushed. If the IV flushes well, then the IV is secured in the usual manner. A secured flushed IV is the definition of a successful IV placement.

Subsequent Attempts:

If unsuccessful with first attempt at IV placement, an attempt at another site with the same technique (VeinViewer™ guided or conventional method) will be performed. This will be repeated until a successful IV is placed or the physician decides to give an alternative therapy that does not need IV access.

We plan to monitor the success rate for DIVA patients who are not enrolled in the study to demonstrate that they are comparable to our control group.

Planned Analysis

VeinViewer™ vs Conventional method:

The main outcome is success or failure of peripheral IV placement on first attempt (a dichotomous outcome). A Chi square test will be used to compare the proportion of subjects with successful first stick IV placement using the VeinViewer™ technique to that using the conventional method with 95% confidence intervals around the difference. Also, planned is to look at the median number of attempts to place IV with each of the different methods of IV placement. We plan to use a non-parametric test like the Wilcoxon Rank sum test. To test for independent associations between VeinViewer™ technique or conventional method for IV placement and success or failure of IV placement on first attempt, multivariate logistic regression will be performed, with potential confounding variables (patient weight, diagnosis, etc) included as co-variates in the model. We plan to use an interaction term in the model that will take in account that there may be a learning curve for the technique (nurses early in the study vs. nurses later in the study).

DIVA score validation:

The patients whose information we collected (validation cohort) in this study will be used to validate the DIVA score. We will determine first attempt success rate with conventional IV placement method at each DIVA score in both the derivation cohort (from data previously collected in the derivation study) and the validation cohort. We will use chi-square statistics to compare derivation and validation cohorts. The areas under the receiver operating characteristics curves for predicting successful IV placement on first attempt at each DIVA score will be compared between the derivation and validation cohorts. Attempts will be made to refine the score should analysis demonstrates that it is warranted.

Estimated sample size calculation: From a previous study, we demonstrated that patients with a DIVA score ≥ 3 had a more than 45% first attempt failure rate for peripheral IV placement using the conventional method. A technique that can improve success by 25% would be considered significant. Using alpha of 0.05, beta of 0.10 (Power = 0.90), and making the question two-tailed; we find an estimated sample size in each group of 85. In other words, 170 children with DIVA ≥ 3 will be needed for our study.

Risk to Subjects:

There are no extra risks expected above that of receiving a standard IV. The standard risks of IV include bleeding, bruising, pain, and infection. The use of the VeinViewer™ technique may or may not take more time to place an IV. If a delay would be detrimental to the subject's care, they will not be asked to take part in this study.

Anticipated significance of the study:

A technique that improves the first stick success rate or decreases the number of sticks required to place an IV would decrease amount of pain, discomfort, and anxiety for the patient. Getting an IV in a timely manner can alter parental perceptions of the quality of care and improve parental satisfaction. Also, this may be a time saver for nurses.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to the emergency department at Children's Hospital of Wisconsin (CHW)
* 0 to 19 years of age
* Requires a peripheral IV as determined by the examining physician
* DIVA score ≥ 3
* During times when VeinViewer™ machine is available
* During hours when a VeinViewer™ trained participating nurse is on duty

Exclusion Criteria:

* Central line available
* Immunocompromised patient
* Requirement for immediate IV placement (Patient's condition would potentially be compromised if there is a time delay in IV placement.)

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
First attempt IV success rates | Immediately after attempt

SECONDARY OUTCOMES:
Number of attempts required | Immediately after attempts

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Yen, MD MS, Principal Investigator — Medical College of WIsconsin and Children's Research Institute; Anne Riegert, RN, Principal Investigator — Children Hospital of Wisconsin Health Systems; Marc H Gorelick, MD MSCE, Principal Investigator — Medical College of Wisconsin and Children's Research Institute
Locations (1):
- Children's Hospital of Wisconsin Emergency Department and Trauma Center, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Yen K, Gorelick MH. Ultrasound applications for the pediatric emergency department: a review of the current literature. Pediatr Emerg Care. 2002 Jun;18(3):226-34. doi: 10.1097/00006565-200206000-00020. No abstract available. PMID 12066016
- [Background] Yen K, Riegert A, Gorelick MH. Derivation of the DIVA score: a clinical prediction rule for the identification of children with difficult intravenous access. Pediatr Emerg Care. 2008 Mar;24(3):143-7. doi: 10.1097/PEC.0b013e3181666f32. PMID 18347490
- [Derived] Abel WM, Efird JT, Crane PB, Ferdinand KC, Foy CG, DeHaven MJ. Use of coaching and technology to improve blood pressure control in Black women with hypertension: Pilot randomized controlled trial study. J Clin Hypertens (Greenwich). 2023 Jan;25(1):95-105. doi: 10.1111/jch.14617. Epub 2022 Dec 20. PMID 36537265
- [Derived] Abel WM, Spikes T, Greer DB. A Qualitative Study: Hypertension Stigma Among Black Women. J Cardiovasc Nurs. 2021 Mar-Apr 01;36(2):96-103. doi: 10.1097/JCN.0000000000000759. PMID 33148961